CLINICAL TRIAL: NCT01180569
Title: Lenalidomide Therapy In Previously Untreated, Advanced Stage Follicular Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-022
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Lymphoma; Follicular Lymphoma
Keywords: Lenalidomide; 10-022
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Lenalidomide

ARMS (1):
- lenalidomide (Experimental): Eligible patients for this clinical trial will be treated for 6 cycles with lenalidomide at 15 mg daily by mouth on Days1-21 of 28 day cycle, preceded by an escalating schema for safety (5mg daily for 2 weeks; 10 mg daily for 2 weeks; and 15 mg daily for 2 weeks) and then a one week rest).
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — Patient enrollment FNA of palpable lymph node prior to escalation phase
  Escalation phase of Lenalidomide:
  Lenalidomide 5 mg daily PO x 14 days Lenalidomide 10 mg daily PO x 14 days Lenalidomide 15 mg daily PO x 14 days Week of rest FNA of palpable lymph node prior to treatment phase
  Treatment phase of Lenalidomide:
  15 mg daily PO days 1-21 out of a 28 day cycle Repeat x 6 cycles

SUMMARY:
The purpose of this study is to see if a treatment with Lenalidomide, which is a pill given by mouth for 7.5 months (30 weeks total), can delay the growth of lymphoma or shrink the lymphoma. Lenalidomide is a pill that has been approved by the Food and Drug Administration (FDA). It is used to treat some forms of cancer-like illnesses (myelodysplastic syndrome (MDS)and in combination with dexamethasone for patients with multiple myeloma (MM) who have received at least 1 prior therapy. MDS and MM are cancers of the blood). This drug works by stimulating the body's immune system and by reducing the blood supply to cancer cells. Cancer cells need blood to live and grow. In this study, the drug is considered a new or experimental drug because we are learning how it works against your form of lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of follicular lymphoma: grades I, II, or IIIA, (as defined in the WHO classification3) as reviewed by a hematopathologist at Memorial Hospital
* No prior treatment for lymphoma permitted.
* Measurable or evaluable disease is permitted; at least one peripheral site amenable to FNAs
* Laboratory test results within these ranges
* Absolute neutrophil count ≥ 2000
* Platelet count ≥ 150,000
* Creatinine clearance of ≥ 60 mL/min (may be actual or calculated by Cockroft-Gault formula
* Total bilirubin 1.5 x ULN
* AST (SGOT) and ALT (SGPT) ≤ 3 x ULN. Karnofsky performance status > 70%
* The patient may not have a previous history of radiation therapy.
* Patient or guardian must be able to sign voluntary written consent.
* Male or female patients 18 years of age or greater.
* Females of childbearing potential (FCBP)† must have a negative serum pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods (Appendix B), and also Appendix C: Education and Counseling Guidance Document.
* Able to take aspirin (81 mg, if not already on aspirin) daily as prophylactic anticoagulation (Patients intolerant to ASA may use low molecular weight heparin). Although not recommended as prophylactic anti-coagulation, warfin may be used with clode monitoring of INR.

Exclusion Criteria:

* Histologic diagnosis of follicular grade 3B or aggressive non-Hodgkin's lymphoma.
* Histologic evidence of transformation from low grade/indolent NHL to aggressive NHL.
* PET uptake in any of the involved sites greater than 12 (suggesting histologic transformation).
* Regional lymphoma (peripheral stages I and II) eligible for involved field irradiation.Staging fulfills criteria for no initial treatment according to GELF criteria2 for advanced stage disease (not peripheral stage I and II amenable to involved field irradiation) . None of the following should be present:

  1. A nodal or extranodal mass with a diameter of >7 cm,
  2. Involvement of at least three nodal sites [each with a diameter of >3 cm],
  3. Systemic symptoms,
  4. Symptomatic splenomegaly, or
  5. Ureteral compression.
* Patients with a known history of HIV, Hepatitis B or C seropositivity.
* Patients with stool positive for H. Pylori (these patients are eligible for protocol 07-038).
* Evidence of laboratory TLS by Cairo-Bishop Definition of Tumor Lysis Syndrome (see Appendix E). Subjects may be enrolled upon correction of electrolyte abnormalities.
* Patients who require therapy with systemic corticosteroids.
* Prior history of malignancy within the past five years or a concurrent malignancy, with the exceptions of cutaneous basal cell carcinoma or carcinoma in situ of the uterine cervix.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Response rate (CR + PR). | 2 years
  The primary objective of this study is to evaluate lenalidomide in previously untreated patients with advanced stage follicular lymphoma who do not require active lymphoma therapy.

SECONDARY OUTCOMES:
Response rate (CR + PR) and time to disease progression | 2 years
  according to FLIPI score. The Follicular Lymphoma International Prognostic Index (FLIPI)
Immune monitoring and analysis of signal transduction in the lymph node. | 2 years
Immune monitoring and analysis of signal transduction in the blood. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Carol Portlock, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm